CLINICAL TRIAL: NCT07341256
Title: Effect of a Short Postpartum Father-Focused Breastfeeding Education on Paternal Support Behaviors and Breastfeeding Outcomes at 1, 3, and 6 Months: A Randomized Controlled Trial
Brief Title: Father-Focused Breastfeeding Education and Breastfeeding Outcomes
Acronym: FBF-EDU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Timuçin İmdadoğlu (Other)
Responsible Party: Sponsor-Investigator, Timuçin İmdadoğlu, Pediatrician, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SVIH-2025-FBF-RCT; EthicsApproval-2025-502 (Other: University of Health Sciences Turkey - Sancaktepe Training and Research Hospital)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Paternal Support; Exclusive Breastfeeding
Keywords: Father-focused breastfeeding education; Paternal involvement; Breastfeeding outcomes; Partner Breastfeeding Influence Scale; Postpartum period
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in parallel to either a father-focused breastfeeding education intervention or a control group receiving routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Father-Focused Breastfeeding Education (Experimental): Fathers receive a brief, structured breastfeeding support education in addition to routine care.
  Interventions: Behavioral: Father-Focused Breastfeeding Education
- Routine Care (No Intervention): Participants receive routine postnatal care without additional breastfeeding education.

INTERVENTIONS:
Behavioral: Father-Focused Breastfeeding Education — A short, face-to-face educational session provided to fathers focusing on practical ways to support breastfeeding.
  Arms: Father-Focused Breastfeeding Education

SUMMARY:
Breastfeeding is recommended as the optimal feeding method for infants during the first six months of life. Support from fathers or partners plays an important role in initiating and maintaining breastfeeding. However, most breastfeeding education programs mainly focus on mothers, and structured education directed to fathers is limited.

This study aims to evaluate the effect of a short, structured, father-focused breastfeeding education given shortly after birth on paternal support behaviors and breastfeeding outcomes. Fathers of healthy term newborns will be randomly assigned to receive either a brief breastfeeding support education or routine care. Paternal support behaviors will be assessed using a validated questionnaire, and infant feeding outcomes will be evaluated during follow-up.

The results of this study may help improve breastfeeding support strategies by involving fathers more actively in the early postnatal period.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized controlled trial conducted at Sancaktepe Prof. Dr. Ilhan Varank Training and Research Hospital in Istanbul, Turkey. The study evaluates the impact of a short, structured, father-focused breastfeeding education delivered in the early postpartum period on paternal breastfeeding support behaviors and infant feeding outcomes.

Fathers or partners of term, clinically stable newborns who are present in the hospital within 24 to 48 hours after birth and who provide written informed consent are eligible for participation. After baseline assessment, participants are randomized in a 1:1 ratio to either the intervention group or the control group.

At baseline, sociodemographic data are collected, and paternal breastfeeding support behavior is assessed using the Turkish version of the Partner Breastfeeding Influence Scale (PBIS-TR). Fathers in the intervention group receive a brief, face-to-face breastfeeding support education lasting approximately 8 to 10 minutes. The education is based on international breastfeeding recommendations and focuses on practical ways fathers can support breastfeeding. The control group receives routine clinical care without additional intervention.

Paternal breastfeeding support behavior is reassessed at one month postpartum. Infant feeding status is evaluated at 1, 3, and 6 months postpartum and categorized as exclusive breastfeeding, partial breastfeeding, or formula/other feeding. Data are analyzed to compare paternal support behaviors and breastfeeding outcomes between the two study groups.

This study aims to provide evidence on the effectiveness of early, father-focused breastfeeding education in improving breastfeeding support and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Fathers or partners aged 18 years or older.
* Fathers or partners of healthy term newborns (≥37 weeks gestation).
* Newborns without major congenital anomalies or chronic medical conditions.
* Fathers or partners present during the early postnatal period.
* Ability to understand and communicate in Turkish.
* Provision of written informed consent.

Exclusion Criteria:

* Fathers or partners of preterm infants (<37 weeks gestation).
* Newborns requiring neonatal intensive care unit admission.
* Newborns with major congenital anomalies or severe medical conditions.
* Fathers or partners unable to complete follow-up assessments.
* Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-03 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Paternal breastfeeding support behavior and exclusive breastfeeding at 1 month postpartum | 1 month postpartum
  Paternal breastfeeding support behavior will be assessed using the Turkish version of the Partner Breastfeeding Influence Scale (PBIS-TR). Infant feeding status at 1 month postpartum will be recorded and categorized as exclusive breastfeeding or non-exclusive breastfeeding.

SECONDARY OUTCOMES:
Infant feeding status at 3 months postpartum | 3 months postpartum
  Infant feeding status will be assessed at 3 months postpartum and categorized as exclusive breastfeeding, partial breastfeeding, or formula/other feeding.
Infant feeding status at 6 months postpartum | 6 months postpartum
  Infant feeding status will be assessed at 6 months postpartum and categorized as exclusive breastfeeding, partial breastfeeding, or formula/other feeding.

CONTACTS AND LOCATIONS:
Overall Officials: timucin imdadoglu, MD, Principal Investigator — University of Health Sciences Turkey, Sancaktepe Prof. Dr. Ilhan Varank Training and Research Hospital
Locations (1):
- Sancaktepe Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rempel LA, Rempel JK. The breastfeeding team: the role of involved fathers in the breastfeeding family. J Hum Lact. 2011 May;27(2):115-21. doi: 10.1177/0890334410390045. Epub 2010 Dec 20. PMID 21173422
- [Background] World Health Organization. Implementation guidance: protecting, promoting and supporting breastfeeding in facilities providing maternity and newborn services - the revised Baby-friendly Hospital Initiative 2018. Geneva: World Health Organization; 2023.